CLINICAL TRIAL: NCT00002225
Title: A Phase II, Open-Label, Multicenter Study to Characterize the Effectiveness and Safety of Efavirenz in Combination With Stavudine and Didanosine in Antiretroviral Therapy-Naive HIV-Infected Patients
Brief Title: A Study of Efavirenz in Combination With Stavudine and Didanosine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dupont Merck (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 281D; DMP 266-044
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; Reverse Transcriptase Inhibitors; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Stavudine; Didanosine

INTERVENTIONS:
Drug: Efavirenz
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give efavirenz plus stavudine plus didanosine to HIV-infected patients who have never received anti-HIV treatment.

DETAILED DESCRIPTION:
Patients will be given combination treatment with efavirenz, stavudine, and didanosine.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection with plasma HIV-RNA greater than or equal to 10,000 copies/ml.
* A life expectancy of at least 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current bilateral peripheral neuropathy greater than or equal to Grade 2.
* Any clinically significant laboratory findings obtained during the screening evaluation (see laboratory values).
* Any clinically significant disease (other than HIV infection) or clinically significant findings during screening of medical history or physical examination.
* Any malignancy that requires systemic therapy.
* Proven or suspected acute hepatitis due to any cause.
* Recurrent episodes of moderate to severe diarrhea, or vomiting lasting more than 4 days within 3 months prior to dosing.
* Active AIDS-defining opportunistic infection or disease.

Concurrent Medication:

Excluded:

Astemizole, cisapride, clarithromycin, ketoconazole, itraconazole, midazolam, rifabutin, rifampin, terfenadine, thalidomide, triazolam, vincristine, zalcitabine.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* Life expectancy less than 12 months.
* Difficulty in swallowing capsules/tablets.
* Hypersensitivity to any component of the formulation of efavirenz, stavudine, or didanosine.

Prior Medication:

Excluded:

* Any other experimental drug within 30 days of introducing study treatment.
* Vaccination within 3 weeks of screening visit.
* Interferon started within 30 days of initiating study treatment.
* Prior antiretroviral therapy.

Risk Behavior:

Excluded:

- Current alcohol or illicit drug use which would interfere with compliance with dosing schedule and protocol evaluations.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Whitman Walker Clinic, Washington D.C., District of Columbia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - North Shore AIDS Hosp / Division of Infectious Disease, Manhassett, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Carolinas Research Associates, Charlotte, North Carolina